CLINICAL TRIAL: NCT02321189
Title: The Effect of Resveratrol Based Nutritional Supplement on Choroidal Thickness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xufang Sun, study director, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: Sun3
Record Dates: First submitted 2014-11-08; First posted 2014-12-22 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Eye Disease
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LONGEVINEX (Placebo Comparator): The Effect of LONGEVINEX on Choroidal Thickness
  Interventions: Drug: LONGEVINEX
- placebo (Placebo Comparator): The Effect of placebo on Choroidal Thickness
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: LONGEVINEX — let everyone of the participants oral 1 capsule containing 100 mg LONGEVINEX
  Arms: LONGEVINEX
Drug: placebo — let everyone of the participants oral 1 capsule containing 100 mg placebo
  Arms: placebo

SUMMARY:
Choroidal thickness represents blood-flowing of eyes. The investigators detect the choroidal thickness of the young participant using SD-OCT to see the effect of Resveratrol Based Nutritional Supplement on Choroidal Thickness.

DETAILED DESCRIPTION:
34 young, healthy participants were included in this study; They were randomly divided into two groups by age and gender matched.100 mg Longevinex® capsule was given to the study group and 100mg placebo capsule to the control group. All participants underwent OCT scanning with spectral domain optic coherence tomography (SD-OCT) at baseline and 1 h following Longevinex® or placebo administration. The choroidal thickness was measured manually by the Heidelberg Eye explore software(version 5.3.3.0, Heidelberg Engineering) with a vertical line to the retinal pigment epithelial layer.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 23-28 years of age. nonsmokers.
2. Patients were considered to be healthy on the basis of electrocardiogram (ECG), and clinical laboratory safety tests (haematology, plasma biochemistry, urinalysis and hepatitis B, hepatitis C and HIV serology) performed at screening.
3. Avoid ingesting grapefruit, grapefruit juice or other grapefruit juice containing products, and any herbal-based nutrient supplement or prescribed medications( grapefruit, cranberry, blueberry products, peanuts and peanut butter, grape and grape products, and red wine ) during the same period of time.
4. patients should abstain from alcohol-containing beverages at least two days prior to and during the study.

Exclusion Criteria:

1. Uncontrolled Blood pressure exceeding diastolic pressure of 100 mm Hg (sitting) during the screening period and uncontrolled diabetes mellitus
2. Participation in another simultaneous medical investigation or trial Renal failure requiring dialysis or renal transplant or liver dysfunction History of other disease,or other findings giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug, might affect interpretation of the results of the study, or render the subject at high risk from treatment complications.
3. IOP over 30 mmHg.
4. Any previous retinal laser photocoagulation to the study eye in treatment naive. Any previous intravitreal injection in study eye (triamcinolone or other) in treatment naive.
5. Any previous vitrectomy in study eye (posterior or anterior associated with vitreous loss in cataract surgery).
6. Intracapsular cataract extraction (posterior capsule needs to be present).
7. Aphakia or absence of the posterior capsule in the study eye, Structural damage to the center of the macula in the study eye preexisting to CRVO likely to preclude improvement in visual acuity following the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s).

Ages: 23 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Choroidal Thickness(micrometer) | baseline
  using Heidelberg Eye Explorer software to measure choroidal thickness of participants

SECONDARY OUTCOMES:
Choroidal Thickness(micrometer) | 1 hour after baseline
  using Heidelberg Eye Explorer software to measure choroidal thickness of participants

CONTACTS AND LOCATIONS:
Overall Officials: Xunfang Sun, Study Director — Department of Ophthalmology,Tongji Hospital, Tongji Medical College, Huazhong University of science and Technology
Locations (1):
- Tongji Medical College of HUST, Wuhan, Hubei, China